CLINICAL TRIAL: NCT00984646
Title: A Single-centre, Placebo- and Standard-care-controlled, Double-blind, Randomised Trial to Investigate the Efficacy of Eight Doses of RN1003 in the Reduction of Scarring From the Approximated Wound Margins of Incisional Wounds
Brief Title: Investigation Into the Scar Reduction Potential of Prevascar (Interleukin-10)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1003-0027
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Wound Healing
Keywords: Cicatrix; Scar; Wound-healing; Prevascar; Interleukin-10 (IL-10); Ilodecakin; RN1003
MeSH Terms: conditions — Cicatrix | interventions — Interleukin-10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal Prevascar (Experimental)
  Interventions: Drug: Prevascar
- Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prevascar — Intradermal Prevascar, 5ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Prevascar — Intradermal Prevascar, 50ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Prevascar — Intradermal Prevascar, 250ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Prevascar — Intradermal Prevascar, 1000ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Prevascar — Intradermal Prevascar, 25ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Prevascar — Intradermal Prevascar, 125ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Prevascar — Intradermal Prevascar, 500ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Prevascar — Intradermal Prevascar, 2000ng/100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Other Names: IL-10; Ilodecakin; RN1003
  Arms: Intradermal Prevascar
Drug: Placebo — Intradermal Placebo, 100μl/linear cm of wound site or margin administered once just prior to wounding and once 24 h later
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study was to investigate the scar-reducing properties of eight doses of intradermal Prevascar (IL-10).

DETAILED DESCRIPTION:
Subjects were randomised to one of two dose groups, each with four concentrations of intradermal Prevascar. Subjects had four 1cm incisional wounds made on the inner aspect of each upper arm (eight in total), giving four sets of anatomically paired wound sites per subject. Each subject acted as their own control with one site from each wound pair randomly treated with intradermal Prevascar and the other treated with Placebo (vehicle) or Standard Care.

Intradermal Prevascar was administered at 100μl per linear cm of wound site prior to wounding on Day 0 and 100μl per linear cm to each wound margin 24 hours later on Day 1. Group 1 subjects received doses of 5, 50, 250 and 1000ng/100μl and group 2 subjects received 25, 125, 500 and 2000ng/100μl.

Subjects in each group were also randomised into two control subgroups to receive either 100μl/linear cm intradermal placebo (Subgroup 1) or Standard Care alone (Subgroup 2) at control wound sites.

Subjects returned for follow-up at Day 14, Month 1, Month 3, Month 6, Month 9 and Month 12.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-85 years, who have given written informed consent
* Subjects with a BMI (Quetelet's index) within the permitted weight/height2 range of 15-55kg/m2
* Subjects with, in the opinion of the Investigator, clinically acceptable results for screening laboratory tests performed within 28 days prior to the first trial administration
* Female subjects with child-bearing potential who are using a method(s) of contraception deemed acceptable by the Investigator and agree to continue doing so for the first month of the trial

Exclusion Criteria:

* Subjects who, on direct questioning and by physical examination, reveal a history or evidence of hypertrophic or keloid scarring
* Subjects with tattoos or previous scars within 3cm of the area to be incised during the trial
* Subjects of Afro-Caribbean descent, because of their increased susceptibility to hypertrophic or keloid scarring
* Subjects who have had previous surgery in the area to be incised, conducted within 1 year of the first dosing day
* Subjects with a history of a bleeding disorder or who are receiving anticoagulant therapy
* Subjects who, on direct questioning and physical examination, show evidence of any past or present clinically significant disease that may affect the endpoints of the trial, e.g. coagulation disorders, diabetes, immuno- mediated conditions and clinically significant skin diseases or allergies
* Subjects with a clinically significant skin disorder that is chronic or currently active, and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial
* Subjects with any clinically significant medical condition or history that would impair wound healing, including significant rheumatoid arthritis, chronic renal impairment (significant for age), significant hepatic impairment (liver function tests >3 times upper limit of normal), congestive heart failure, active malignancy or history of malignancy within last 5 years, immunosuppression or chemotherapy within last 12 months, history of radiotherapy or diabetes mellitus
* Subjects with a history of hypersensitivity to any of the drugs or dressings used in the trial
* Subjects who are taking, or who have taken, any investigational product or participated in a clinical trial within 3 months prior to the first trial
* dose administration
* Subjects who are taking regular, continuous, oral corticosteroid therapy
* Subjects undergoing investigations or changes in management for an existing medical condition
* Subjects with a history of drug abuse, or who test positive for drugs of abuse (cocaine, amphetamines, methamphetamines, opiates or benzodiazepines) during the screening period, which is not explained by the intake of legitimate prescribed or over-the-counter medication for a documented medical condition
* Subjects who, in the opinion of the Investigator, are unlikely to complete the trial for whatever reason
* Subjects receiving immunosuppressive treatment
* Females who are pregnant or lactating
* Subjects who have any clinically significant neurological impairment or disease
* Subjects with an active infection (subjects were able to participate in the trial once the infection had passed and they had been re-screened)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2005-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To establish which of eight intradermal doses of RN1003 has the greatest scar-reducing properties, compared with Placebo and Standard Care. | 12 months

SECONDARY OUTCOMES:
To collect further safety and tolerability data for RN1003 | 12 months
To assess pre- and post-dose systemic levels of RN1003. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James Bush, Principal Investigator — Renovo
Locations (1):
- Renovo, Manchester, United Kingdom

REFERENCES:
- [Derived] Do NN, Willenborg S, Eckes B, Jungst C, Sengle G, Zaucke F, Eming SA. Myeloid Cell-Restricted STAT3 Signaling Controls a Cell-Autonomous Antifibrotic Repair Program. J Immunol. 2018 Jul 15;201(2):663-674. doi: 10.4049/jimmunol.1701791. Epub 2018 Jun 13. PMID 29898959